CLINICAL TRIAL: NCT01240005
Title: A Phase I/II Evaluation of Cytokine Induced Killer Cells Stimulated by DC(DCIK) Immunotherapy in Patients With Renal Cell Carcinoma
Brief Title: Cytokine Induced Killer Cells Stimulated by DC Immunotherapy for Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: An Yongheng,Li Yanjiang,Gao Hong,Zhang Xuefeng, The Affilited Hospital of Medical College,Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCCIK002
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCIK (Experimental)
  Interventions: Biological: DCIK

INTERVENTIONS:
Biological: DCIK — Renal cell carcinoma patients were treated with three intravenous infusions of DC activated CIK cells at 1-day intervals. Clinical examinations of these patients were performed.

SUMMARY:
30% of renal cell carcinoma patients have metastases, mostly in lung, liver and bones at the time of diagnosis. Because of poor response to radiation therapy or chemotherapy, several studies have been initiated to find alternative therapeutic options.

Cytokine induced killer cells(CIK) are an unique population of cytotoxic T lymphocytes with a characteristic CD3+ CD56+ phenotype; they can be generated from cytokine cocktail-induced peripheral blood mononuclear cells (PBMC). CIK cells represent strong anti-tumor cytotoxicity in vitro and in vivo. Interestingly,the anti-tumor activity of CIK cells can be enhanced by incubation with dendritic cells (DC), which are the most potent antigen (Ag)-presenting cells.

The purpose of this study was to evaluate the clinical efficacy of DC-activated CIK cell treatment following regular therapy and the effects of this therapy on immune responses in patients with renal cell carcinoma after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, adult patients of 18 to 75 years of age at time of diagnosis that qualify for standard treatment including surgery.
2. Histologically confirmed diagnosis of renal cell carcinoma.
3. Newly diagnosed or recurrent disease.
4. Karnofsky performance status 60-100.
5. Life expectancy ≥ 12 weeks.
6. Written informed consent of patient and/or legal guardian.
7. Must be off steroid at least two weeks prior to vaccination.
8. Hematologic and metabolic panel results will be within the parameters of the protocol.
9. Normal renal function in the kidney.
10. Adequate function of liver,lung and heart.
11. Negative pregnancy test
12. Fertile patients must use effective contraception
13. Serologically negative for HIV,HBV,HCV.
14. Syphilis serology negative
15. Patient must have no prior sensitivity to the components of the dendritic cell vaccine.

Exclusion Criteria:

1. Anti-neoplastic chemotherapy or radiotherapy during 4 weeks before entering the study.
2. Presence of acute infection.
3. Inability to obtain informed consent because of psychiatric or complicating medical problems.
4. Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
5. Subjects with organ allografts.
6. Known history of autoimmune disorder.
7. Pregnancy or breast-feeding.
8. Positive for hepatitis B, C, HIV, syphilis.
9. Patients unwilling to perform a save method of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year

SECONDARY OUTCOMES:
Objective tumor response, Time to recurrence, Progression-free, Cellular immunity. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yongheng An, Study Chair — The affilited hospital of medical college,Qingdao university
Locations (1):
- Stem cell cencter of the affiliated hospital of medical colledge,qingdao university, Qingdao, Shandong, China